CLINICAL TRIAL: NCT00849342
Title: A Prospective, Multicentre, Non-controlled, Observational, 52-weeks Study: the Evaluation of the Body Weight Progress During the Treatment With Insulin Detemir in Type 1 or 2 Diabetes Patients, Previously Treated With Other Basal Insulins
Brief Title: Observational Study on Levemir® in Obese Diabetic Patients
Acronym: KILOS
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN304-3708
Record Dates: First submitted 2009-02-20; First posted 2009-02-23 (Estimated); Last update posted 2014-08-15 (Estimated); Status verified 2014-07

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2 | interventions — Insulin Detemir

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A
  Interventions: Drug: insulin detemir

INTERVENTIONS:
Drug: insulin detemir — Safety and effectiveness (weight and HbA1c) data collection in connection with the use of the drug Levemir® in daily clinical practice.

SUMMARY:
This study is conducted in Europe. The aim of this observational study is to investigate the effect of switch from other basal insulin treatments to Levemir® on body weight in obese diabetic patients. A local extension will be conducted in Slovenia in order to reach the planned 400 patients for the sub-analysis of Slovenian patients.

Included in the study is a retrospective part to evaluate the weight progress since initiation of insulin treatment of another basal insulin and/or oral antidiabetic drugs (OAD) and/or bolus insulin therapy. Retrospective data will be collected at baseline and at approximately 6 and 12 months before starting insulin detemir therapy.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes mellitus (Type 1 or type 2)
* BMI greater than 27 kg/m^2, or more than 3 kg weight increase since start of insulin therapy

Exclusion Criteria:

* Subjects currently being treated with insulin detemir
* Subjects who were previously enrolled in this study;
* Subjects with a hypersensitivity to insulin detemir or to any of the excipients.
* Women who are pregnant, breast feeding or have the intention of becoming pregnant within next 12 months Female patients will be reminded to use adequate contraceptive during the study, where is relevant.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients from both general and speciality practice settings who have been deemed appropriate to receive Levemir® because of weight increase on other insulin therapies, and as part of routine out-patient care by the prescribing physician.
Sampling Method: Non-Probability Sample
Enrollment: 580 (Actual)
Dates: Start 2008-12; Primary Completion 2011-04 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Change in body weight and BMI | during 12 months of treatment

SECONDARY OUTCOMES:
Change in body weight at different BMI subgroups | at insulin start, 12 and 6 months before treatment and after 3, 6, 9 and 12 months of treatment
Change in waist perimeter | from insulin start and after 6 and 12 months of treatment
Change in FPG (Fasting Plasma Glucose) | from 12 and 6 months before treatment after 6 and 12 months of treatment
Change in HbA1C | from insulin start and 12 and 6 months before treatment and after 6 and 12 months of treatment
Change in number of hypoglycaemic events during 4 weeks proceeding routine visits | after 6 and 12 months of treatment
Number of adverse drug reactions (ADR) | after 6 and 12 months of treatment
Change in blood pressure | from insulin start and 6 and 12 months after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (2):
- Alphen aan den Rijn, Netherlands
- Ljubljana, Slovenia

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com